CLINICAL TRIAL: NCT04767412
Title: Improvement of Physical Fitness by Inspiratory Muscle Training in Children With Down Syndrome
Brief Title: Inspiratory Muscle Training and Physical Fitness in Children With Down Syndrome Randomized Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reham Saeed Alsakhawi, Assistant Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/ 012/001922
Record Dates: First submitted 2021-02-19; First posted 2021-02-23 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Down Syndrome
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aerobic exercise (Active Comparator)
  Interventions: Device: aerobic exercise training, inspiratory muscle training
- aerobic exercise and inspiratory muscle training (Active Comparator)
  Interventions: Device: aerobic exercise training, inspiratory muscle training

INTERVENTIONS:
Device: aerobic exercise training, inspiratory muscle training — All participants received 30 min of aerobic exercise training thrice per week for a period of 12 weeks, whereas the group B received an additional 30 min of IMT before each aerobic exercise session.

SUMMARY:
The purpose of this study is to investigate the effect of inspiratory muscle training on physical fitness in Down syndrome children. Twenty Down syndrome children from both genders ranged in age chronologically from seven to ten years will be selected to participate in this study. Selection of the study sample and evaluation of physical fitness improvement as well as Inspiratory Muscle training will be conducted in the Down Syndrome Charitable Association (DSCA), Riyadh City.

The study sample will be divided randomly into two equal groups of (A & B). All the children participated in the current study will receive 30 minutes of treatment session of aerobic exercise, group B will receive first 30 minutes of IMT then take a period time of rest about 30 minutes before starting the aerobic exercise. Exercise frequency three times per week for a period of three successive months.

The Body mass index (BMI) of each participated child will be determined by measuring weight/ Kg and height/ m2 using Electronic weight and height scale to include BMI ≥ 29 Kg/ m2 to exclude the obese children. Also using Six Minute Walk Test (6MWT) for measuring the aerobic capacity and Pulse Oxymeter for measuring pulse rate and Oxygen saturation. In addition, The Gio Digital pressure gauge will be used to assess Respiratory Muscle Strength of children by determining the Maximal Inspiratory (MIP) and Expiratory Pressure (MEP) which used to detect the inspiratory training intensity and reflect the improvement in respiratory muscle strength after training program. Brockport Physical Fitness Test (BPFT) will be used to measure physical fitness of the participated children. The participated children will be assessed before and after three successive months .

The obtained results of this study will measure Maximal Inspiratory (MIP) and Expiratory Pressure (MEP), Aerobic capacity, Musculoskeletal Function and Maximum Heart Rate (HR Max.) to determine the significant improvement of participated children

ELIGIBILITY:
Inclusion Criteria:

* children with a body mass index (BMI) ≥ 25 kg/m2, and
* children with the ability to understand and follow verbal commands and instructions used during training and tests

Exclusion Criteria:

* with neurological, visual, or auditory defect,
* with asthma or any chronic chest diseases,
* with significant tightness or deformities in the lower limbs,
* with obesity, or
* who performed regular physical activity

Ages: 10 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2021-01-21 (Actual)

PRIMARY OUTCOMES:
maximal inspiratory pressure | 2 months

SECONDARY OUTCOMES:
maximal expiratory pressure | 2 months
aerobic capacity | 2 months
endurance | 2 months
  using the 6MWT

CONTACTS AND LOCATIONS:
Overall Officials: Reham Alsakhawi, Ph.D, Principal Investigator — Assistant Professor, Faculty of Physical Therapy, Cairo University
Locations (1):
- Faculty of Physical Therapy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Elshafey MA, Alsakhawi RS. Inspiratory Muscle Training and Physical Fitness in Children With Down Syndrome: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2022 Dec;103(12):2279-2287. doi: 10.1016/j.apmr.2022.04.005. Epub 2022 May 6. PMID 35533737